CLINICAL TRIAL: NCT05788718
Title: A Multicenter, Prospective, Observational Study to Analyze the Prescription Pattern of Sugammadex and Its Effectiveness and Safety in Non-interventional, Real-world Setting
Brief Title: An Observational Study to Analyze the Prescription Pattern of Sugammadex and Its Effectiveness and Safety
Acronym: SECURE
Status: Completed | Type: Observational
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: BR-SGD-OS-401
Record Dates: First submitted 2023-02-09; First posted 2023-03-29 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Complications; Neuromuscular Blockade; Anesthesia
Keywords: sugammadex; rocuronium; vecuronium
MeSH Terms: conditions — Postoperative Complications | interventions — Sugammadex

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Sugammadex — As this is a non-interventional study designed to collect data as part of routine clinical practice, the type and dose of neuromuscular blocking agents are all based on the clinician's judgment.

SUMMARY:
The purpose of this observational study is to evaluate patients who are planning to administer sugammadex after rocuronium or vecuronium is used.

The main questions it aims to answer are:

1. Prescription pattern of sugammadex
2. Effectiveness and safety of sugammadex

Since this study is observational, only data generated under daily treatment are to be collected, and no additional tests or drug administration is conducted for the study. The patients are observed from baseline to 24 hours after the initial administration of sugammadex.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults aged 19 or older
* Is to undergo elective surgery under general anesthesia
* Is planned to use rocuronium or vecuronium as an NMBA
* Is planned for extubation before/after being moved to the recovery room
* ASA physical status I - III
* Patients who have signed the informed consent after receiving information about the purpose and method of this study

Exclusion Criteria:

* Has myasthenia gravis or Eaton-Lambert myasthenic syndrome
* Has hypersensitivity to ingredients of sugammadex, rocuronium, or vecuronium
* Has received an investigational product within 12 weeks from the study enrollment or has plans to participate in another clinical trial during the participation of this study.
* Other subjects who are considered inappropriate to participate in this study by the judgment of the investigator.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are planning to undergo surgery using rocuronium or vecuronium for the neuromuscular blockade and planned to receive sugammadex for the antagonist.
Sampling Method: Non-Probability Sample
Enrollment: 6458 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-05-08 (Actual)

PRIMARY OUTCOMES:
Re-administration rate of sugammadex | baseline~24 hours after administration
  The number and ratio of patients re-administered with sugammadex within 24 hours of the initial administration of sugammadex are evaluated.

SECONDARY OUTCOMES:
Prescription pattern of sugammadex | baseline~24 hours after administration
  The ratio of patients is presented for each administered time and dose.
Incidence rate of postoperative residual curarization (PORC)(TOFr<0.9) | at 3 and 30 minutes after administration of sugammadex
  The TOFr (train-of-four ratio) is measured at 3 and 30 minutes after administration of sugammadex. The number and ratio of patients with a TOFr <0.9 are defined as PORC(TOFr<0.9). The TOFr is expressed as a decimal from 0.0 up to 1.0.
Incidence rate of postoperative residual curarization (PORC)(TOFr<1.0) | at 3 and 30 minutes after administration of sugammadex
  The TOFr (train-of-four ratio) is measured at 3 and 30 minutes after administration of sugammadex. The number and ratio of patients with a TOFr <1.0 are defined as PORC(TOFr<1.0). The TOFr is expressed as a decimal from 0.0 up to 1.0.
Analysis of clinical factors affecting sugammadex re-administration | baseline~24 hours after administration
  The number and ratio of patients who had these clinical factors are evaluated.
Incidence rate of respiratory complications related to postoperative residual muscle relaxation after surgery | time from the first administration of sugammadex ~ 24 hours after administration
  The number and ratio of patients who had respiratory complications related to postoperative residual muscle relaxation after surgery are evaluated.
TOFr before sugammadex administration | baseline~24 hours after administration
  The TOFr (train-of-four ratio) is measured before each administration of sugammadex. The TOFr is expressed as a decimal from 0.0 up to 1.0.
TOFr before extubation | baseline~24 hours after administration
  The TOFr (train-of-four ratio) is measured before extubation. The TOFr is expressed as a decimal from 0.0 up to 1.0.
Time to extubation | baseline~24 hours after administration
  The time from the first administration of sugammadex or the last administration of NMBA to the time of extubation is measured in minutes.
Time surpassed from the expected dismissal time from the recovery room | baseline~24 hours after administration
  The time of dismissal from the recovery room is recorded for each patient.
Ratio of unplanned transfer to the intensive care unit(excluding lung surgery and heart surgery) | time from the first administration of sugammadex ~ 24 hours after administration
  The number and ratio of patients who was moved from the recovery room to the intensive care unit unplanned.
Incidence rate of PONV(postoperative nausea and vomiting) | time from the first administration of sugammadex ~ 24 hours after administration
  The number and ratio of patients who experiences PONV(postoperative nausea and vomiting).
Incidence rate of adverse drug reaction | time from the first administration of sugammadex ~ 24 hours after administration
  The number and ratio of patients who experiences adverse drug reactions in which their relationship to sugammadex cannot be ruled out.
Incidence rate of serious adverse drug reaction | time from the first administration of sugammadex ~ 24 hours after administration
  The number and ratio of patients who experiences serious adverse drug reactions in which their relationship to sugammadex cannot be ruled out.

CONTACTS AND LOCATIONS:
Overall Officials: Choon-Hak Lim, MD, Principal Investigator — Department of Anesthesiology and Pain Medicine, Korea University Medical Center, Seoul, Korea.
Locations (1):
- Korea University Anam Hospital, Seoul, Seongbuk-gu, South Korea

IPD SHARING:
Plan to Share IPD: No